CLINICAL TRIAL: NCT01432587
Title: The Effect of Diflunisal on Familial Transthyretin Amyloidosis: An Open Label Extension Study of "the Diflunisal Trial" (IND 68092), and an Open Label Observational Study on Previously Untreated Patients With Familial Transthyretin Amyloidosis.
Brief Title: The Effect of Diflunisal on Familial Transthyretin Amyloidosis
Acronym: DFNS01
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Ole B Suhr, Professor, MD, PhD, Professor MD PhD, Umeå University
Other Study IDs: DFNS01; 2011-000776-34 (EudraCT Number)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; Transthyretin; Neuropathies; Diflunisal; Familial
MeSH Terms: conditions — Amyloidosis | interventions — Diflunisal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Whole blood Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Diflunisal — Film-coated tablet, 250 mg twice daily, orally for approximately 2 years

SUMMARY:
An ongoing trial of diflunisal has been closed for enrollment, thus, patients suitable for the study can no longer participate or receive treatment by diflunisal; and patients, who have participated in the trial can not continue their treatment. The investigators want to continue to monitor the effect of the drug on transthyretin (TTR) amyloidosis in an open label observational study.

Primary endpoint will be a composite score of the manifestations of the disease (Kumamoto scale) and secondary end points will be measurements of neurological impairment, heart involvement and nutritional status.

DETAILED DESCRIPTION:
Duration of treatment in this study is dependent of the results from the ongoing IND 68092-study, which are planned to be presented 2013.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy and genetically proven systemic transthyretin amyloidosis caused by a TTR gene mutation. The amyloid shall be proven to be of transthyretin type, and the fibril composition settled.
* Age ≥ 18 years.
* Negative pregnancy test and contraception for sexually active women of child bearing potential.

Exclusion Criteria:

* Concomitant use of non-study non-steroidal anti-inflammatory drugs (NSAIDs)
* Heart failure with symptoms at daily activities (NYHA class ≥III)
* Renal insufficiency (creatinine clearance < 30 ml calculated from the Cockcroft-Gault formula)
* Active non-haemorrhoidal bleeding within the last 18 month.
* Non-treated peptic ulcer disease.
* Anticoagulation therapy, low dose ASA permitted.
* Non-steroidal or aspirin allergy/hypersensitivity
* Thrombocytopenia (< 100,000 platelets/mm3)
* Inability or unwillingness of subject to give written informed consent
* By the investigator regarded as unable to follow the study guidelines and scheduled controls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting the Units for Familal amyloidosis in Umeå, Piteå and Skellefteå
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in the Kumamoto scale | Enrollment, 12 month and annual follow-up
  Composite score of the manifestations of the disease (Kumamoto Scale). Results at enrollment will be compared to results at 12 months and annual follow-ups.

SECONDARY OUTCOMES:
Changes in modified body mass index (mBMI) | Enrollment, 12 month and annual follow-up
  Changes in nutritional status measured by mBMI.Results at enrollment will be compared to results at 12 months and annual follow-ups.
Changes in paraneoplastic neurological disorders (PND) scale | Enrollment, 12 month and annual follow-up
  Neurological impairment measured by the PND-score. Results at enrollment will be compared to results at 12 months and annual follow-ups.
Changes in cardiac function | Enrollment, 1 month, 2 month, 3 month, 6 month, 9 month 12 month, 18 month and annual follow-up
  Cardiac impairment is measure by echocardiographic measurement of septal thickness and by proBNP in blood samples. Results at enrollment will be compared to results during the study and annual follow-ups.
Safety follow-up Blood Work | 1 month, 3 month, 6 month, 9 month, 12 month and follow-up every 6 months
  To follow-up the patient safety during the study and follow-up the blood samples for (B-Hb), blood platelets, s-creatinine, liver enzymes [aspartate transaminase (ASAT),alanine aminotransferase (ALAT), s-bilirubin and alkaline phosphatase (ALP)],serum proBNP (S-proBNP) are drawn. Results at enrollment will be compares to results during study and every 6-month follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Ole B Suhr, MD PhD, Principal Investigator — Dept of Clinical Medicine and public Health, Umeå University
Locations (3):
- Sweden (3):
  - Dept of Clinical Medicin, Ptieå Hospital, Piteå
  - Dept of clinical medicin, Skellefteå Hospital, Skellefteå
  - Dept of Clinical Medicine, Umeå University Hospital, Umeå